CLINICAL TRIAL: NCT02762305
Title: The Effects of the RSVP Bone Builders Program on Intrinsic Fall Risk Factors & Life Satisfaction
Brief Title: The Effects of the RSVP Bone Builders Program on Strength, Balance, Fall Risk and Life Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Northridge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1516-091
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Exercise
Keywords: fall risk; RSVP bone builders; group exercise; older adults; balance confidence; life satisfaction; balance; walking speed
MeSH Terms: conditions — Motor Activity; Personal Satisfaction

ARMS (1):
- RSVP Bone Builder group exercise (Experimental): A group of older adults who are participating in the RSVP Bone Builder group exercise.
  Interventions: Other: RSVP Bone Builders Group Exercise

INTERVENTIONS:
Other: RSVP Bone Builders Group Exercise

SUMMARY:
The hypothesis of this study is that participation in the Retired and Senior Volunteer Program (RSVP) Bone Builders program 1 hour, twice per week, for 12 weeks may result in significant positive changes to the health status of older adult participants as demonstrated by increased leg strength and walking speed, improved balance and balance confidence, and enhanced life satisfaction. These improvements may lead to a reduction in risk of falls.

DETAILED DESCRIPTION:
The purpose of this study was to examine the efficacy of the RSVP Bone Builders program, to document benefits this program may have for older adults and also provide additional evidence that further confirms the importance of exercise for the older adult population. Exercise has the potential to reduce falls, injuries, emergency room visits, surgeries, insurance costs, and improve the overall quality of life in the older adult population. If the RSVP Bone Builders proves to be beneficial for older adults, the program could be recommended by healthcare and exercise professionals for their patients and clients who are at risk for falls.

ELIGIBILITY:
Inclusion Criteria:

* able to walk independently with or without a cane or walker,
* not currently participating in the RSVP Bone Builders program,
* scoring at least 24/30 on the Mini-Mental State Examination (MMSE) and clearance of Physical Activity Readiness Questionnaire (Par-Q)

Exclusion Criteria:

* if they use a wheelchair in the community for mobility,
* have any known neurological, musculoskeletal, cardiopulmonary, or other medical condition that will not allow full participation in the RSVP Bone Builders program, and
* if the subjects score less than 24/30 on the MMSE

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
10 Meter Walking Test | 12 weeks
  Measures gait speed
Timed Up and Go Test | 12 weeks
  Measures gait speed & fall risk
Five Time Sit to Stand Test | 12 weeks
  Measures leg strength & fall risk
Computerized Dynamic Posturography with NeuroCom Smart Equitest | 12 weeks
  Measures balance abilities & fall risk
Berg Balance Scale | 12 weeks
  Measures balance abilities & fall risk
Activities-specific Balance Confidence (ABC) Scale | 12 weeks
  Measures balance confidence & fall risk
Satisfaction with Life Scale | 12 weeks
  Measures life satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Giannini, Principal Investigator — California State University, Northridge
Locations (1):
- Equilibrium Balance Performance Center, Ventura, California, United States